CLINICAL TRIAL: NCT01963676
Title: Clinical Trial to Assess Transcranial Current Stimulation as a Treatment for Medication Refractory Auditory Hallucinations in Schizophrenia
Brief Title: Transcranial Current Stimulation as a Treatment for Auditory Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Flavio Frohlich, PhD, Assistant Professor, Departments of Psychiatry, Cell Biology and Physiology, and Biomedical Engineering, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-2995
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Auditory Hallucinations
Keywords: schizophrenia; auditory hallucinations; transcranial stimulation; tDCS; tACS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (tDCS) (Experimental): 13 subjects total. 2mA stimulation for 20 minutes.
  Interventions: Device: tDCS
- Sham stimulation (Sham Comparator): 13 subjects total. An initial 40sec of stimulation at 2mA followed by a small current pulse every 550msec for the remainder of the 20 minute period.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: tDCS
  Arms: transcranial direct current stimulation (tDCS)
Device: Sham stimulation
  Arms: Sham stimulation

SUMMARY:
Investigating the effect of non-invasive transcranial current stimulation on auditory hallucinations in patients with schizophrenia. Normal neuronal activity is perturbed in schizophrenia, so selective targeting of this abnormal activity could serve as a treatment for schizophrenia and alleviate symptoms caused by abnormal neuronal activity, such as auditory hallucinations.

DETAILED DESCRIPTION:
AIM 1: To evaluate the effect of transcranial direct current stimulation (tDCS) (2mA for 20min on five consecutive days) on auditory hallucinations in schizophrenia patients using the change in ratings on the Auditory Hallucination Rating Scale (AHRS) by patients before and after stimulation. We hypothesize that tDCS will modulate the abnormal neuronal activity found in schizophrenic patients and thereby decrease their auditory hallucinations when measured after stimulation.

AIM 2: To evaluate the long term effects of tDCS by having patients give a rating on the AHRS after one month has passed since stimulation and comparing this value to their baseline score and their score immediately after stimulation. We hypothesize that there will remain a significant reduction in auditory hallucination score in participants who received tDCS at one month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual IV (DSM-IV) diagnosis of schizophrenia, any subtype, or schizoaffective disorder, with refractory auditory hallucinations. Duration of illness >1 year.
* 18-99 years old.
* Clinically stable for at least 12 weeks, i.e. not requiring hospitalization or a change in level of care .
* On current antipsychotic doses for approximately 4 weeks or more.
* Capacity to understand all relevant risks and potential benefits of the study (informed consent) OR has a legal guardian who can complete consent forms on the patients behalf
* Right handed

Exclusion Criteria:

* Subjects with a DSM-IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months.
* History of significant head injury/trauma, as defined by loss of consciousness for more than 1 hour, or recurring seizures, or requiring later cognitive rehabilitation or causing cognitive sequelae.
* Prior brain surgery.
* Any brain devices/implants, including cochlear implants and aneurysm clips.
* Co-morbid neurological condition (i.e. seizure disorder, brain tumor).
* Medical or neurological illness (unstable cardiac disease AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation.
* Non English speakers.
* Pregnancy, nursing, or if female and fertile, unwilling to use appropriate birth control measures during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Psychiatry
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Outpatient STEP Clinic, Chapel Hill, North Carolina
  - University of North Carolina, Wake STEP Clinic, Raleigh, North Carolina

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited through medical providers. Providers knew inclusion/exclusion criteria and discussed the study with patients during their regular appointments. Interested participants contacted the study team. Participants recruited from the STEP clinic (Chapel Hill and Raleigh), and the Burlington ACT team. Recruitment between 4/14 and 9/14.
Pre-assignment Details: Subjects randomly assigned to one of two groups, transcranial direct stimulation (tDCS) group or active sham group. tDCS group, direct current was delivered during awake, resting state for 20minutes on 5 consecutive days. Sham stimulation was delivered for an equal period of time and number of sessions. 27 subjects signed consent, 1 withdrew.
Groups:
- Transcranial Direct Current Stimulation (tDCS): 13 subjects total. 2mA stimulation for 20 minutes.
  tDCS
- Sham Stimulation: 13 subjects total. An initial 40sec of stimulation at 2mA followed by a small current pulse every 550msec for the remainder of the 20 minute period.
  Sham stimulation
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Stimulation
Started | 14 | 13
Completed | 13 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Based on our randomized block design model, a block size of 10 (subjects, 20 total), 2 levels of (within-factors) TREATMENT and TIME each and a residual standard deviation of 14 (Brunelin et al., 2012), the power of our study is estimated to be 0.85 at the significant level alpha=0.05 and the difference of percentage change in 5 days of 15.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Stimulation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.38 (12.64) | 40.00 (10.74) | 41.69 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Auditory Hallucination Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Remission according to AHRS: AHRS score equal to 0. AHRS: standardized, clinician-administered rating scale; assesses 11 aspects characteristically associated with auditory hallucination. Individual items are scored on a 5 point (0 to 4), with 0=none/absent and 4=most severe. Total score: 0 to 44; higher score indicates more severe auditory hallucination symptoms. Scores for each question summed up for total score.
  units on a scale | 27.00 (6.90) | 26.69 (6.30) | 26.85 (6.48)
Positive and Negative Syndrome Scale [Mean (Standard Deviation); unit: units on a scale] — Remission according to PANSS: PANSS score equal to 30. PANSS: standardized, clinician-administered rating scale. 3 subscales; Positive Symptom scale: 7 items, Negative Symptom scale: 7 items, General Symptom scale: 16 items. Each item in each subscale are scored on a 7 point (1 to 7) scale, with 1=none/absent and 7=most severe. Total score for Positive Scale: 7 to 49. Total score for Negative Scale: 7 to 49. Total score for general scale: 16 to 112. Total score for PANSS: 30 to 210; higher score indicates more severe symptoms. The PANSS total score by adding the sums of each subscale.
  units on a scale | 73.15 (12.90) | 66.92 (17.17) | 70.04 (15.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Auditory Hallucination Rating Scale (AHRS)Score From Baseline to Day 5
Description: Examining AHRS total score after 5 days of stimulation compared to baseline assessment total.
Time Frame: Baseline, Day 5
Population: Per protocol; All participants who completed every session of the study from the initial session through the one month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Stimulation
Number analyzed (Participants) | 13 | 13
units on a scale | -6.38 (6.38) | -8.54 (8.68)
Statistical Analysis 1: Comparison: Transcranial Direct Current Stimulation (tDCS) vs Sham Stimulation; The null hypothesis was that there is no difference between the changes in the AHRS score from baseline to 5 days between the groups: H0: μ1 = μ2 μ1: mean(difference 5 days-baseline) for tDCS group (n=13) μ2: mean(difference 5 days-baseline) for sham group (n=13); Test type: Superiority or Other; p = 0.48, t-test, 2 sided — There was no adjustment because we just performed one comparison; Difference from Day 5 to Baseline was compared between the sham and the tDCS group using an unpaired t-test. Degrees of freedom: df = 24

2. Secondary Outcome: Persistence of Decrease in AHRS Score Over Time
Description: We will re-assess patients one month after the completion of stimulation to evaluate whether their change from baseline to day 5 score on the AHRS persisted over time, namely 30 days.
Time Frame: Day 5, One month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Stimulation
Number analyzed (Participants) | 13 | 13
units on a scale | -5.38 (9.06) | -4.77 (8.26)
Statistical Analysis 1: Comparison: Transcranial Direct Current Stimulation (tDCS) vs Sham Stimulation; The null hypothesis was that there is no difference between the AHRS score changes from baseline to 1month between the groups: H0: μ1 = μ2 μ1: mean(difference 1 month-baseline) for tDCS group (n=13) μ2: mean(difference 1 month-baseline) for sham group (n=13); Test type: Superiority or Other; p = 0.86, t-test, 2 sided — There was no adjustment because we just performed one comparison; Difference from 1 Month to Baseline was compared between the sham and the tDCS group using an unpaired t-test. Degrees of freedom: df = 24

ADVERSE EVENTS:
Time Frame: Adverse event data collected from the beginning of the study (4/2014) through the completion of the study (10/2014) for a total of 6 months.
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No